CLINICAL TRIAL: NCT00101296
Title: Phase I Trial of R115777 (NSC 702818) in Relapsed, Refractory or High Risk Myeloid Leukemia
Brief Title: Tipifarnib in Treating Patients With Relapsed or Refractory Acute Myeloid Leukemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-03078; PHI-47; U01CA062505 (NIH); CDR0000404151 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2005-01-07; First posted 2005-01-10 (Estimated); Last update posted 2013-02-04 (Estimated); Status verified 2013-01

CONDITIONS: Acute Myeloid Leukemia With Multilineage Dysplasia Following Myelodysplastic Syndrome; Adult Acute Erythroid Leukemia (M6); Adult Acute Megakaryoblastic Leukemia (M7); Adult Acute Minimally Differentiated Myeloid Leukemia (M0); Adult Acute Monoblastic Leukemia (M5a); Adult Acute Monoblastic Leukemia and Acute Monocytic Leukemia (M5); Adult Acute Monocytic Leukemia (M5b); Adult Acute Myeloblastic Leukemia With Maturation (M2); Adult Acute Myeloblastic Leukemia Without Maturation (M1); Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Del(5q); Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); Adult Acute Myelomonocytic Leukemia (M4); Adult Erythroleukemia (M6a); Adult Pure Erythroid Leukemia (M6b); Recurrent Adult Acute Myeloid Leukemia; Untreated Adult Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Erythroblastic, Acute; Leukemia, Megakaryoblastic, Acute; Leukemia, Monocytic, Acute; Leukemia, Myeloid, Acute; Congenital Abnormalities; Leukemia, Myelomonocytic, Acute | interventions — tipifarnib

ARMS (1):
- Treatment (tipifarnib) (Experimental): Patients receive oral tipifarnib twice daily on days 1-7 and 15-21. Courses repeat every 28 days in the absence of unacceptable toxicity or disease progression. Patients achieving a CR receive 2 additional courses beyond CR. Patients experiencing relapse after previously achieving CR may receive additional tipifarnib at the current dose level for newly registered patients.
  Interventions: Drug: tipifarnib; Other: pharmacological study; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: tipifarnib — Given orally
  Other Names: R115777; Zarnestra
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
Tipifarnib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. This phase I trial is studying the side effects and best dose of tipifarnib in treating patients with relapsed or refractory acute myeloid leukemia

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To define the maximum tolerated dose (MTD) of R115777 (tipifarnib) in patients with relapsed, refractory, or high risk myeloid leukemias treated according to this regimen.

II. To assess the toxicity and preliminary assessment of efficacy of R115777 in patients with relapsed, refractory, or high risk myeloid leukemias.

OUTLINE: This is a dose-escalation, multicenter study.

Patients receive oral tipifarnib twice daily on days 1-7 and 15-21. Courses repeat every 28 days in the absence of unacceptable toxicity or disease progression. Patients achieving a complete response (CR) receive 2 additional courses beyond CR. Patients experiencing relapse after previously achieving CR may receive additional tipifarnib at the current dose level for newly registered patients.

Cohorts of 3-6 patients receive escalating doses of tipifarnib until the MTD is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

Patients are followed every 6 months for survival.

PROJECTED ACCRUAL: A total of 20-30 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with acute myeloid leukemia (AML), excluding the M3 subtype (acute promyelocytic leukemia), that are not likely to respond to conventional therapy, including:

  * Relapsed or refractory AML after one to three prior induction regimens (not counting consolidation therapies while in CR, such as autologous transplant),
  * Newly diagnosed AML in patients up to age-70 with poor risk features (unfavorable cytogenetics or findings suggestive of prior myelodysplasia) not fit for standard induction therapy, and
  * Newly diagnosed AML patients age 70 - 75 not fit for standard therapy (without history of prior myelodysplastic syndrome [MDS])
* Bone marrow and peripheral blood studies must be available for confirmation of diagnosis; cytogenetics, flow cytometry, and molecular studies (such as fms-related tyrosine kinase 3 [Flt-3] status) will be obtained as per standard practice
* Patients with active central nervous system (CNS) leukemia are NOT eligible
* Performance status of 60% or greater by the Karnofsky scale
* If induction chemotherapy has been attempted, a minimum of 4 weeks must have elapsed since the completion of prior chemotherapy in order to be eligible for this study; hydroxyurea for control of blasts is not counted as chemotherapy, and may be given up until 24 hours before starting R115777
* Patients may have had prior autologous transplant; they must be at least 100 days post transplant, and have had recovery of their counts with ANC > 1000 and platelets greater than 100K at some point post transplant, and be without active CMV or fungal disease
* Patients may have received prior radiation therapy as part of a transplant conditioning regimen; radiotherapy must have been completed at least 100 days prior to starting on R115777
* There are no minimum hematological parameter requirements prior to the first two cycles of R115777, as patients with AML and MDS are understood to have low ANC and platelet counts when the disease is active; however, patients with WBC greater than 30,000 will receive hydroxyurea to reduce WBC to below 30,000 at which point they may begin treatment with R115777
* A pretreatment calculated creatinine clearance (absolute value) of >= 60 ml/minute or serum creatinine of < 1.5 x upper limit of normal is required
* Serum bilirubin =< 2.0 mg/dl
* SGOT and SGPT =< 2.5 times the institutional upper limits of normal
* Any condition causing inability to swallow pills given by mouth will render patients ineligible for the trial
* There must be no plans for the patient to receive concurrent hormonal, biologic, or radiation therapy
* Patients eligible, at the time of starting the drug, for curative therapeutic approaches (such as allogeneic transplant) are not eligible for the trial; however, patients who achieve CR or PR as a result of R115777 may go on to allogeneic transplant
* Patients must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional and federal guidelines
* Prior to the first patient registration, the notification of institutional review board approval for this study must be provided to the Data Coordinating Center at City of Hope
* Antacids are allowed but must not be taken concurrently with R115777; (there must be at least 2 hours between antacid intake and R115777 dosing)
* Pregnant or lactating women are excluded from this trial; all patients of child-bearing potential, both male and female, must be advised to practice adequate contraception; premenopausal women must have a negative pregnancy test prior to entry on this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2004-10; Primary Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
MTD defined as the highest dose level in which six patients have been evaluated for toxicity with no more than one patient experiencing dose limiting toxicity (DLT) assessed using Common Terminology Criteria for Adverse Events (CTCAE) version 3.0 | 28 days
  The toxicities observed at each dose level will be summarized in terms of type, severity, time of onset, duration, and reversibility or outcome. Tables will be created to summarize these toxicities and side effects by dose and by course.
Objective tumor response | Up to 6.5 years
  Will be summarized at each dose level, and the number and percent responding combined across dose levels.
Survival | From registration to time of death due to any cause, assessed up to 6.5 years
  Will be summarized with Kaplan-Meier plots.
Time to treatment failure | From registration to the first observation of disease progression, death due to any cause, or early discontinuation of treatment, assessed up to 6.5 years
  Will be summarized with Kaplan-Meier plots.
Duration of response | Up to 6.5 years
  Will be summarized with Kaplan-Meier plots.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Kirschbaum, Principal Investigator — City of Hope Medical Center
Locations (1):
- City of Hope, Duarte, California, United States